CLINICAL TRIAL: NCT03458260
Title: A Multicentre, Phase II, Open Label, Single Arm Study of Pixantrone in Patients With CD20-positive Relapsed or Refractory Aggressive Non-Hodgkin Lymphoma Treated With Rituximab, Ifosfamide and Etoposide.
Brief Title: Study of Pixantrone in CD20+ Relapsed/Refractory Aggressive Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIVeR
Record Dates: First submitted 2018-02-26; First posted 2018-03-08 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Aggressive Non-Hodgkin Lymphoma
Keywords: Diffuse Large B-Cell Lymphoma (DLBCL); relapsed or refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Recurrence | interventions — pixantrone; Ifosfamide; Etoposide; Rituximab; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Pixantrone plus rituximab, ifosfamide and etoposide.
  Interventions: Drug: Pixantrone; Other: Ifosfamide; Other: Etoposide; Other: Rituximab; Procedure: Transplant

INTERVENTIONS:
Drug: Pixantrone — 6 cycles - dose = 80mg/m²
  Other Names: Pixuvri
Other: Ifosfamide — 6 cycles - 1500 mg/m2
  Other Names: Holoxan
Other: Etoposide — 6 cycles - 150 mg/m2
  Other Names: Vepeside
Other: Rituximab — 6 cycles - 375 mg/m2
  Other Names: Mabthera
Procedure: Transplant — after 2 or 6 cycles

SUMMARY:
This study will evaluate the efficacy of Pixantrone with rituximab, ifosfamide and etoposide as measured by the overall metabolic response rate after 2 cycles of treatment or at permanent treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven CD20+ aggressive non-Hodgkin lymphoma (diffuse large B-cell lymphoma (DLBCL), de novo or transformed DLBCL from previously untreated low grade non-Hodgkin lymphoma or grade 3b follicular lymphoma) as per the World Health Organization (WHO) 2016 criteria
2. Relapsed or refractory disease, defined as follows:

   1. Patients eligible for ASCT who failed to achieve a Complete Response (CR) after at least one salvage therapy (eg, Rituximab-Etoposide- Methylprednisolone - Cytarabine - Cisplatin (R-ESHAP) or Rituximab- Dexamethasone- High-dose Cytarabine - Cisplatin (R-DHAP), patients who were previously refractory to Rituximab-Ifosfamide-Cytarabine-Etoposide (R-ICE) (stable disease or progressive disease) are not eligible to the study)
   2. Or patients in first relapse after Autologous Stem Cell Transplant (ASCT)
   3. Or patients not eligible for ASCT who failed to achieve a CR after at least one prior treatment (and no more than 4 previous lines) or in relapse after at least one prior treatment (and no more than 4 previous lines).
3. Age > or =18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status < or = 2
5. Subjects must have evaluable disease based on positron emission tomography (PET-CT) scan
6. Minimum life expectancy of 6 months
7. Signed written informed consent
8. Patient covered by any social security system
9. Men must agree to use a barrier method of contraception during the treatment period and until 6 months after the last dose of chemotherapy
10. Women of childbearing potential must agree to use an adequate method of contraception, such as oral contraceptives, intrauterine device, or barrier method of contraception during the treatment period and until 12 months after the last dose of chemotherapy

Exclusion Criteria:

1. Any other histological type of lymphoma (Burkitt lymphoma, mantle-cell lymphoma…)
2. Any history of previously treated indolent non-Hodgkin lymphoma
3. Symptomatic central nervous system or meningeal involvement by the lymphoma
4. Contraindication to any drug contained in the Pixantrone with rituximab, ifosfamide and etoposide regimen
5. Treatment with any investigational drug within 28 days before the first study drug administration
6. Any of the following lab abnormalities unless related to the lymphoma or bone marrow infiltration:

   1. Absolute neutrophil count (ANC) < 1.0 G/L
   2. Platelet count < 100 G/L
   3. Creatinine clearance < 40 mL/min for patients < 70 y, or creatinine clearance < 60 mL/min for patients > or = 70 y, by Modification of Diet in Renal Disease (MDRD) method.
   4. Total bilirubin level > 1,5 x Upper Limit of Normal (ULN)
   5. Serum ASpartate Transaminase (AST) or ALanine Transaminase (ALT)> 2,5x ULN
7. Known Human Immunodeficiency Virus (HIV) positive
8. Active hepatitis C virus (HCV) (Positive HCV serology with positive Polymerase Chain Reaction (PCR) for HCV RNA)
9. Active hepatitis B (HB) :

   1. HBsAg positive
   2. HBsAg negative, Ac anti-HBs positive and/or Ac anti-HB core (HBc) positive (Patients who are seropositive due to a history of hepatitis B vaccine are eligible. Patients with Ac anti-HBs positive and/or Ac anti-HBc positive and no history of hepatitis B vaccine are eligible only if PCR for HB virus DNA is negative)
10. Cumulative dose of doxorubicine or equivalent > 450mg/m2
11. Left ventricular ejection fraction (LVEF) < 50% measured by echocardiography or isotopic method
12. Congestive heart failure (any stage from New York Heart Association (NYHA) classification)
13. Uncontrolled arterial hypertension
14. Severe rhythmic heart disease
15. Uncontrolled ischemic heart disease, including patients with stable angina
16. Significant valvular heart disease
17. History of a myocardial infarction within 6 months prior to enrolment
18. Pregnant or lactating females
19. Prior history of malignancies with the exception of non-melanoma skin tumors (basal cell or squamous cell carcinoma) or in situ cervical carcinoma
20. Any serious active disease or co-morbid medical condition according to the investigator's decision
21. Adult person unable to provide informed consent because of intellectual impairment, any serious medical condition, laboratory abnormality or psychiatric illness
22. Use of any standard or experimental anti-cancer drug therapy within 28 days before the first study drug administration
23. Use of corticosteroids prior to baseline PET-CT
24. Person deprived of his/her liberty by a judicial or administrative decision
25. Person hospitalized without consent
26. Adult person under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Overall Metabolic Response rate (OMR) according to local investigator | After 42 days of treatment (2 cycles) or at permanent treatment discontinuation.
  by local investigator according to Lugano classification 2014

SECONDARY OUTCOMES:
Complete Metabolic Response rate (CMR) according to local investigator | After 42 days of treatment (2 cycles of 21 days) or at permanent treatment discontinuation.
  according to local investigator
Overall Metabolic Response rate (OMR) according to central review | After 42 days of treatment (2 cycles of 21 days) or at permanent treatment discontinuation.
  according to local investigator
Complete Metabolic Response rate (CMR) according to central review | After 42 days of treatment (2 cycles of 21 days) or at permanent treatment discontinuation.
  according to local investigator
Number of Adverse Events (AEs) and Serious Adverse Events (SAEs) | After 42 or 126 days of treatment (2 or 6 cycles of 21 days) or at permanent treatment discontinuation.
Number of patients for whom Partial Metabolic Response (PMR) is transformed into CMR | After 42 days of treatment (2 cycles of 21 days) or at permanent treatment discontinuation.
Rate of ASCT | After 42 days of treatment (2 cycles of 21 days) or at permanent treatment discontinuation.
  Number of patients who perform an ASCT out of total number of patients
Success of stem cell collection after treatment | After 42 days of treatment (2 cycles of 21 days) or at permanent treatment discontinuation.
  Rate of successful stem cell collection

CONTACTS AND LOCATIONS:
Overall Officials: Luc-Matthieu Fornecker, Principal Investigator — CHU de Strasbourg; Eric Van den Neste, Principal Investigator — UCL St Luc Bruxelles; Sandy Amorin, Principal Investigator — Hôpital St Louis - Paris
Locations (22):
- Belgium (3):
  - AZ Sint Jan, Bruges
  - Institut Jules Bordet - Centre des tumeurs de l'ULB, Brussels
  - Centre Hospitalier de Jolimont, Haine-Saint-Paul
- France (19):
  - CH d'Avignon, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHU Jean Minjoz, Besançon
  - Hôpital Haut-Lévèque, Bordeaux
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - Clinique Victor Hugo, Le Mans
  - CHRU de Lille, Lille
  - CHU Lyon Sud, Lyon
  - CHU de la Conception, Marseille
  - Centre Lacassagne, Nice
  - Hopital La Pitié Salpétriere, Paris
  - Hôpital St louis, Paris
  - CHU de Poitiers, Poitiers
  - Centre Hospitalier Annecy Genevois, Pringy
  - CH de Cornouaille, Quimper
  - Hôpital Robert Debré, Reims
  - CHU de Rouen, Rouen
  - CHU de Strasbourg, Strasbourg
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No